CLINICAL TRIAL: NCT05929833
Title: A Randomized Controlled Trial of BETTER, A Transitional Care Intervention, for Patients With Traumatic Brain Injury and Their Families
Brief Title: BETTER (Brain Injury Education, Training, and Therapy to Enhance Recovery)
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00112309
Record Dates: First submitted 2023-04-14; First posted 2023-07-03 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-10

CONDITIONS: Traumatic Brain Injury
Keywords: transitional care; patients; family caregivers
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BETTER TBI (Traumatic Brain Injury) Transitional Care Intervention (Experimental): Skilled clinical interventionists follow a manualized intervention protocol to address patient/family needs; establish goals; coordinate post-hospital care, services, and resources; and provide patient/family education and training on self- and family-management and coping skills <16 weeks post-discharge.
  Interventions: Behavioral: BETTER (Brain Injury, Education, Training, and Therapy to Enhance Recovery)
- Usual Care (Placebo Comparator): In alignment with U.S. usual care for patients with TBI (Traumatic Brain Injury), usual care arm activities for younger adults with TBI and their family caregivers will includes usual care discharge planning process and follow up (e.g., verbal and written discharge instructions, with guidance on medications, outpatient therapy, and follow-up appointments).
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: BETTER (Brain Injury, Education, Training, and Therapy to Enhance Recovery) — The six components of BETTER include: 1) assessment of patient/family needs and referral to community-based resources; 2) patient goal setting and review of goals; 3) health care coordination; 4) availability of clinical interventionist to patient/family; 5) training on self- and family-management and brain injury coping skills; and 6) warm hand off/referral to the state-affiliated Brain Injury Association at the end of the intervention for additional resources.
  Arms: BETTER TBI (Traumatic Brain Injury) Transitional Care Intervention
Other: Usual Care — Usual care discharge planning process and follow up (e.g., verbal and written discharge instructions, with guidance on medications, outpatient therapy, and follow-up appointments)
  Arms: Usual Care

SUMMARY:
Despite poor outcomes for adults with traumatic brain injury (TBI), there are no U.S. standards for TBI transitional care for patients discharged home from acute hospital care. To enhance the standard of care, we will examine the efficacy of our existing intervention named BETTER (Brain Injury, Education, Training, and Therapy to Enhance Recovery), a patient- and family-centered TBI transitional care intervention, compared to usual care, among adults with TBI and families. The knowledge generated will drive improvements in outcomes for adults with TBI and families, resulting in improved health of the public.

DETAILED DESCRIPTION:
Patients with TBI (age 18 and older) with mild-to-severe traumatic brain injury (TBI) face high incidence and hospitalization rates, and poor cognitive, physical, behavioral, and emotional impairments <12 months post-discharge. These impairments affect patients' abilities to independently manage their health, wellness, and activities of daily living, resulting in dependence on family. The complexity of needs combined with the fragmentation of healthcare services creates the perfect storm for low patient quality of life (QOL), mismanaged symptoms, rehospitalizations, and increased caregiver strain. Lack of insurance or access to care aggravate these ongoing issues. Despite complex health needs, there are no U.S. standards for transitional care for patients with TBI. Transitional care is defined as actions in the clinical encounter designed to ensure the coordination and continuity of healthcare for patients transferring between different locations or levels of care (e.g., acute hospital care to home). In other patient groups with acute events (e.g., stroke, myocardial infarction), transitional care interventions have led to improved patient QOL and health outcomes. Yet, few TBI transitional care interventions exist. The paucity of theory-driven, evidence-based TBI transitional care interventions led our team to develop an intervention named BETTER (Brain Injury, Education, Training, and Therapy to Enhance Recovery). Based on the Individual and Family Self-Management Theory (IFSMT), BETTER is a patient- and family-centered, behavioral intervention for adults with TBI discharged home from acute hospital care and families. The goal is to improve patients' QOL (change in SF-36 total score, primary outcome) by 16-weeks post-discharge, as this timeframe includes high rates of unmet patient/family needs and preventable clinical events. Skilled clinical interventionists follow a manualized intervention protocol to address patient/family needs; establish goals; coordinate post-hospital care, services, and resources; and provide patient/family education and training on self- and family-management and coping skills <16 weeks post-discharge. Findings from our NIH R03 pilot study showed BETTER significantly improved patients' physical QOL by 31.36 points (p = 0.006) and that the intervention was feasible and acceptable with adults with TBI and families. Thus, the purpose of this study is to examine the efficacy of BETTER (vs. usual care) among adults with TBI who are discharged home from acute hospital care and families. Findings will guide our team in designing a future, multi-site trial to disseminate and implement BETTER into clinical practice to ultimately drive advancements to enhance the standard of care for adults with TBI and families.

ELIGIBILITY:
Patients with TBI, regardless of insurance status, will be eligible if they are/have:

* age 18 years or older;
* diagnosed with mild, moderate, or severe TBI [admission Glasgow Coma Scale score of 3-15];
* admitted to a Duke University Hospital inpatient acute care unit;
* plans to be discharged directly home from Duke University Hospital without inpatient rehabilitation or transfer to other settings (community discharge);
* sufficient cognitive functioning to participate (i.e., able to follow 2-step commands), as determined by the Galveston Orientation and Amnesia Test (score >76 eligible);
* English- or Spanish-speaking (self-report);
* access to a phone or computer with internet capabilities for study participation

Patients with TBI will be excluded if they have/are:

1. Pre-injury neurologic conditions/disorder(s):

   The following neurological conditions/disorders are excluded:

   • untreated ADHD, cerebral palsy, stroke, multiple sclerosis, Parkinson's disease); pre-injury cognitive impairments (e.g., Alzheimer's disease and related dementias); and developmental disorders (e.g., autism, down's syndrome).

   The following neurological conditions are not being excluded:

   • transient ischemic attack, small vessel disease; essential tremor; concussion (maximum 2 prior concussions with no prior history of post-concussion syndrome); myasthenia gravis; dysautonomia; foot drop; degenerative disc disease; spine reticulopathy; bell's palsy + other cranial nerve palsy; neurogenic bladder (if in isolation); and epilepsy [patients with epilepsy are eligible to participate if they had no hospital admissions or emergency department visit for seizures in the last 6 months]
2. Severe psychiatric diagnosis (i.e., untreated schizophrenia, untreated bipolar 1 or 2, any indication of psychosis or acute psychotic events occurring) that are untreated with no psychiatric provider on record, which would preclude patients from having capacity to consent
3. Admitted from settings or locations other than home
4. No family caregiver to participate

Family members will include patient-identified biological relatives and friends and are eligible if they are/have:

* associated with a patient meets all above-listed patient criteria;
* age 18 years or older;
* an anticipated primary caregiver after discharge (i.e., plans to live in same home as patient or have direct contact with patient >10 hours/week);
* English- or Spanish-speaking (self-report);
* access to a phone or computer with internet capabilities for study participation.

Family members will be excluded if the associated patient is not eligible or declines participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-01-26 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in patient SF-36 (36-item Short Form Survey) score | baseline (24-72 hours pre-discharge); 8-, 16-, and 24-weeks post-discharge
  The SF-36 is a quality of life (QOL) measurement with a score range of 0 to 100, where a higher score indicates a better outcome.

SECONDARY OUTCOMES:
Change in patient cognitive function (Neuro-QOL, Cognitive functioning) | baseline (24-72 hours pre-discharge); 8-, 16-, and 24-weeks post-discharge
  The Neuro-QOL is a self-report of health related quality of life for individuals with neurological disorders. Raw scores are converted to T-scores with a mean of 50 and standard deviation of 10.
Change in patient physical functioning (Neuro-QOL, Upper & Lower extremity functioning) | baseline (24-72 hours pre-discharge); 8-, 16-, and 24-weeks post-discharge
  The Neuro-QOL is a self-report of health related quality of life for individuals with neurological disorders. Raw scores are converted to T-scores with a mean of 50 and standard deviation of 10.
Change in patient sleep disturbance (NeuroQOL Sleep Disturbance, short-form) | baseline (24-72 hours pre-discharge); 8-, 16-, and 24-weeks post-discharge
  The Neuro-QOL is a self-report of health related quality of life for individuals with neurological disorders. Raw scores are converted to T-scores with a mean of 50 and standard deviation of 10.
Change in patient TBI-related symptoms (Rivermead Post-concussion questionnaire) | baseline (24-72 hours pre-discharge); 8-, 16-, and 24-weeks post-discharge
  The Rivermead Post-concussion questionnaire is a self-reported measures of TBI-related symptoms. Scores on the first 3 items of the RPQ can range from 0 to 12, with higher scores indicated higher severity of early symptom clusters of post-concussive symptoms; scores on items 4 to 16 can range from 0 to 52, with higher scores indicating higher severity of later post-concussive symptoms
Change in patient participation [Participation Assessment with Recombined Tools-Objective (PART-O)] | 8-, 16-, and 24-weeks post-discharge
  Participation will be measured using the Participation Assessment with Recombined Tools-Objective (PART-O), an objective measure of societal participation developed for patients with TBI with 24-items, with higher scores indicating higher levels of participation
Change in patient process of care transition [Care Transitions Measure-3 (CTM-3)] | 8-, 16-, and 24-weeks post-discharge
  The process of care transitions will be measured by the Care Transitions Measure-3, a 3-item scale with scores ranging from 0 to 100, with higher scores indicating less challenges with the transitional care process
Change in patient and caregiver difficulty accessing services [Service Obstacles Scale (SOS)] | 8-, 16-, and 24-weeks post-discharge
  Difficulty accessing services will be measured by the Service Obstacles Scale, a 6-item scale with scores ranging from 7 to 42, with higher scores indicating more difficulty accessing services
Change in patient and caregiver quality of life / health status (Euro Qol, 5 Item [EQ-5D-5L]) + VAS (visual analog scale) + Cognitive domain (C) | baseline (24-72 hours pre-discharge); 8-, 16-, and 24-weeks post-discharge
  The EQ-5D-5L is a patient reported outcome consisting of 5 items asking about quality of life. EQ-5D-5L index scores range from -0.59 to 1, where 1 is the best possible health state. The VAS (visual analog scale) captures self-rated health. Patients with TBI will also complete the cognitive domain of the EuroQol (EQ-5D-5L+C), to capture condition specific issues, but caregivers will not.
Change in patient and caregiver multi-dimensional interpersonal processes of care in the clinical encounter [Interpersonal Processes of Care (IPC) short-form] | baseline (24-72 hours pre-discharge); 8-, 16-, and 24-weeks post-discharge
  Multi-dimensional interpersonal processes in the clinical encounter, particularly discrimination in the clinical encounter, will be measured using the Interpersonal Processes of Care survey (short-form). The measure, which contains 18-items, has 7 domains using a 1 to 5 scale, with scores ranging from 18 to 90. Higher scores indicate a higher frequency of interpersonal challenges and discrimination in the clinical encounter.
Change in patient and caregiver depressive symptoms [PHQ-9 (Patient Health Questionnaire-9)] | baseline (24-72 hours pre-discharge); 8-, 16-, and 24-weeks post-discharge
  The PHQ-9 assesses degree of depression severity via questionnaire. It has a score range of 0 to 27, where a higher score indicates greater depression.
Change in patient and caregiver Self-Efficacy for Management of Chronic Conditions Scale | baseline (24-72 hours pre-discharge); 8-, 16-, and 24-weeks post-discharge
  The Self-Efficacy to Manage Chronic Disease Scale is made up of 6 items on a visual analog scale, ranging from 1 (not at all confident) to 10 (totally confident). The total score range is 6 to 60, where a higher score indicates greater confidence.
Change in patient and caregiver alcohol and substance abuse (CAGE-AID Substance Abuse Screening Tool) | baseline (24-72 hours pre-discharge); 8-, 16-, and 24-weeks post-discharge
  Alcohol and substance use will be measured using the CAGE-AID Substance Use Screening Tool, a 5-item measure with scores ranging from 0 to 4, with higher scores indicating higher possibility of substance use disorder and need for possible testing
Score on patient and family personal health literacy (Self-Reported Health Literacy Questions) | baseline (24-72 hours pre-discharge)
  Health literacy will be measured using the Self-Reported Health Literacy Questions, a 3-item measure with scores ranging from 3-15, with higher scores indicating lower self-reported health literacy.
Number and type of healthcare services utilized | 8-, 16-, and 24-weeks post-discharge
  Measured by patient and/or caregiver proxy report of patient transitional health care utilization, using a survey developed by the team.
Change in caregiver Modified Caregiver Strain Index (MCSI) | baseline (24-72 hours pre-discharge); 8-, 16-, and 24-weeks post-discharge
  The MCSI can quickly screen for caregiver strain in long-term caregivers. Scoring is 2 points for each 'yes', 1 point for each 'sometimes', and 0 for each 'no' response. The total score ranges from 0 to 26, where a higher score indicates a higher level of caregiver strain.
Change in caregiver Preparedness for Caregiving Scale | baseline (24-72 hours pre-discharge); 8-, 16-, and 24-weeks post-discharge
  The Preparedness for Caregiving Scale is a caregiver self-rated instrument that consists of eight items that asks caregivers how well prepared they believe they are for multiple domains of caregiving. Responses are rated on a 5 point scale with scores ranging from 0 (not at all prepared) to 4 (very well prepared). The scale is scored by calculating the mean of all items answered with a score range of 0 to 4. The higher the score the more prepared the caregiver feels for caregiving.
Score on Pittsburgh Rehabilitation Participation Scale (PRPS) | weekly from 1- to 16-weeks post-discharge
  The interventionist/transitional care manager will rate the patient and the caregiver on the Pittsburgh Rehabilitation Participation Scale (PRPS) to capture their level of engagement in Brain Injury Coping Skills (BICS) sessions. The PRPS is a clinician-rated instrument designed to assess a patient's participation in therapy. The PRPS will only be used for treatment arm participants.
Time spent caregiving and caregiving responsibilities | baseline (24-72 hours pre-discharge); 8-, 16-, and 24-weeks post-discharge
  Time spent caregiving and caregiving responsibilities will be measured using 3 items created by the study team.
Change in Patient Activation Measure (PAM-10) for patients and caregivers. | baseline (24-72 hours pre-discharge); 8-, 16-, and 24-weeks post-discharge
  The Patient Activation measure will that assesses a patient's and caregiver's ability to manage their health and healthcare. Insignia Health's proprietary survey scoring algorithm produces a PAM Score along an empirical, interval-level scale from 0-100 that correlates to one of four levels of patient activation. PAM Levels 1 and 2 indicate lower patient activation, while PAM Levels 3 and 4 indicate higher patient activation.

OTHER OUTCOMES:
Demographics | baseline (24-72 hours pre-discharge)
  Age, sex, race/ethnicity, education, pre-injury occupation, insurance status, annual income
Clinical Factors | baseline (24-72 hours pre-discharge)
  TBI severity, length of stay, comorbidities (via chart review)

CONTACTS AND LOCATIONS:
Overall Officials: Tolu O Oyesanya, PhD, RN, Principal Investigator — Duke University School of Nursing
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
The proposed research will involve a sample of approximately N=500 individuals recruited from Duke University Hospital, located in Durham, NC. The final dataset will include self-reported demographic data, data collection measures, information recorded from study interventionists, and qualitative interview data (audio recordings and transcripts). We will be collecting identifying information. Although the final dataset will be de-identified, we believe there remains the possibility of deductive disclosure of participants with unusual characteristics. Thus, we will make data and associated documentation available to users only under a data-sharing agreement that provides for a commitment to: 1) using de-identified data only for research purposes and not to identify any individual participant; 2) securing the data using appropriate computer technology; and 3) destroying or returning the data after analyses are completed.

REFERENCES:
- [Background] Oyesanya TO, Ibemere SO, You H, Emerson MM, Pan W, Palipana A, Kandel M, Ingram D, Soto M, Pioppo A, Albert B, Walker-Atwater T, Hawes J, Komisarow J, Ramos K, Byom L, Gonzalez-Guarda R, Van Houtven CH, Agarwal S, Prvu Bettger J. Efficacy of BETTER transitional care intervention for diverse patients with traumatic brain injury and their families: Study protocol of a randomized controlled trial. PLoS One. 2024 Feb 23;19(2):e0296083. doi: 10.1371/journal.pone.0296083. eCollection 2024. PMID 38394279
- See also: Efficacy of BETTER transitional care intervention for diverse patients with traumatic brain injury and their families: Study protocol of a randomized controlled trial — https://pubmed.ncbi.nlm.nih.gov/38394279/